CLINICAL TRIAL: NCT07054060
Title: Endarterectomy Versus Stenting in Patients With Symptomatic Severe Carotid Stenosis - 2
Acronym: EVA3S-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D24-P001; PHRC-22-0121 (Other Grant/Funding Number: Ministry of health, France); 2024-A01377-40 (Other: GHU Paris)
Record Dates: First submitted 2025-05-13; First posted 2025-07-08 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: CEA, CAS; stroke; Magnetic resonance imaging; Carotid Artery Stenting; Carotid Endarterectomy
MeSH Terms: conditions — Stroke; Apraxias | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgical arm (Active Comparator): carotid endarterectomy
  Interventions: Procedure: carotid endarterectomy
- Stenting arm (Active Comparator): Carotid artery stenting
  Interventions: Procedure: Carotid artery stenting

INTERVENTIONS:
Procedure: carotid endarterectomy — Carotid endarterectomy is a surgical procedure used to reduce the risk of stroke due to carotid artery stenosis. During an endarterectomy, the surgeon opens the artery and removes the plaque.
  Arms: surgical arm
Procedure: Carotid artery stenting — Carotid artery stenting is an endovascular procedure in which a stent is deployed in the lumen of the carotid artery to treat narrowing of the carotid artery and reduce the risk of stroke.
  Arms: Stenting arm

SUMMARY:
Carotid stenosis caused by atherosclerosis is a significant risk factor for ischemic stroke, accounting for up to 15% of all strokes and transient ischemic attacks. Randomized clinical trials (RCTs) have demonstrated the benefits of carotid endarterectomy (CEA) in reducing stroke risk in patients with severe symptomatic carotid stenosis. Carotid artery stenting (CAS) has been developed as an alternative to CEA, offering several potential advantages, such as avoiding local surgical complications. However, unlike CEA, CAS has not been compared to medical therapy in RCTs for symptomatic carotid stenosis.

DETAILED DESCRIPTION:
CEA vs CAS Comparison:

Early RCTs conducted in the 2000s showed that CAS was associated with a higher risk of procedural stroke or death compared to CEA (8.9% vs 5.8%; RR 1.53, 95% CI 1.20-1.96, p=0.0006). However, CAS was found to be as effective as CEA in preventing recurrent ipsilateral strokes up to 10 years after treatment. Interestingly, an ancillary study of the ICSS trial showed that significantly more patients in the CAS group (50%) than in the CEA group (17%) had new ischemic lesions on diffusion-weighted MRI (DWI), suggesting that DWI might serve as a surrogate outcome measure for future carotid intervention trials.

Data Analysis and Recent Advances:

Individual pooled data analysis of RCTs indicated that CAS could be as safe and effective as CEA in patients under 70 years old. Recent advances in CAS technology, stenting techniques, antiplatelet therapy, and pre-treatment imaging have improved the periprocedural safety of CAS. Due to its ability to treat patients soon after a stroke, CAS has become increasingly used in routine clinical practice.

Study Objectives:

The question remains whether CAS is as safe as CEA in patients with recent symptomatic severe carotid stenosis. The study's objectives are:

Primary Objective:

To assess whether carotid stenting is non-inferior to carotid endarterectomy in preventing new ischemic lesions on DWI MRI, confirmed by a core lab.

* To assess the difference between groups regarding post-intervention MRI characteristics in terms of ischemic lesion number and size, vessel occlusion and hemorrhagic transformation
* To assess differences between groups with regard to the procedural risks and efficacy (within 30 days after procedure) of

  1. any stroke or death
  2. any stroke,
  3. disabling or fatal stroke
  4. death
  5. transient ischemic attack
  6. myocardial infarction
  7. local complication
  8. cranial nerve palsy

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years or over
* Hemispheric or retinal transient ischemic attack or a non-disabling stroke (or retinal infarct) within 15 days before enrolment
* Stenosis of 50% to 99% in the symptomatic carotid artery (NASCET method) for whom revascularisation is decided according to guidelines

Exclusion Criteria:

* Patients unwilling or unable to participate in follow-up for whatever reason
* Preexisting disability (Modified Rankin Score ≥ 3)
* Nonatherosclerotic carotid disease
* Severe tandem lesions
* Previous revascularization of the symptomatic carotid stenosis
* History of bleeding disorder
* Unstable angina
* Contraindication to dual antiplatelet therapy
* Contraindication to MRI
* Life expectancy of less than 2 years
* Percutaneaous or surgical intervention within 30 days before or after the study procedure
* Stenotic lesion on arterial workup appeared as not a factor in the selection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2028-03-16 (Estimated); Study Completion 2028-03-16 (Estimated)

PRIMARY OUTCOMES:
DWI Lesion Detection Rate | From 3 days before procedure to 7 days after procedure
  Imaging endpoint : Proportion of patients having at least one new lesion on post-treatment Diffusion-Weigthed Imaging (DWI) MRI compared to pre-treatment DWI MRI and confirmed by a core lab.
  The pre-treatment DWI MRI will be performed within 3 days before procedure. The post-treatment DWI MRI will be performed within 7 days after procedure.

SECONDARY OUTCOMES:
Profile of lesions | From 3 days before procedure to 7 days after procedure
  Imaging endpoint : Number and size of new lesions on post-treatment MRI. The pre-treatment DWI MRI will be performed within 3 days before procedure. The post-treatment DWI MRI will be performed within 7 days after procedure.
Vessel Occlusion Profile | From 3 days before procedure to 7 days after procedure
  Imaging endpoint : Proportion of patients having a new intracranial vessel occlusion on post-treatment MRI.
  The pre-treatment DWI MRI will be performed within 3 days before procedure. The post-treatment DWI MRI will be performed within 7 days after procedure.
Hemorrhage | From 3 days before procedure to 7 days after procedure
  Imaging endpoint : Hemorrhagic transformation on post-treatment MRI. The pre-treatment DWI MRI will be performed within 3 days before procedure. The post-treatment DWI MRI will be performed within 7 days after procedure.
Stroke/Mortality | From randomization to 30 days after procedure
  Clinical endpoint : proportion of patients having any stroke or death during periprocedural period.
Stroke Incidence Rate | From randomization to 30 days after procedure
  Clinical endpoint : Proportion of patients having any stroke during periprocedural period.
Severe Stroke Incidence | From randomization to 30 days after procedure
  Clinical endpoint : Proportion of patients having any disabling or fatal stroke during periprocedural period.
Mortality | From randomization to 30 days after procedure
  Clinical endpoint : Proportion of patients who died during periprocedural period.
TIA Incidence | From randomization to 30 days after procedure
  Clinical endpoint : Proportion of patients having a Transient ischemic attack during periprocedural period.
MI Occurrence | From randomization to 30 days after procedure
  Clinical endpoint : Proportion of patients having myocardial infarction during periprocedural period.
Local complication | From randomization to 30 days after procedure
  Clinical endpoint : cervical or groin or radial hematoma, infection, arteriovenous fistula at puncture site, lower-limb arterial occlusion during periprocedural period.
Cranial Nerve Injury Events | From randomization to 30 days after procedure
  Clinical endpoint : Proportion of patients having cranial nerve injury during periprocedural period.
Hospitalization Duration | From the date of the carotid artery stenting (CAS) or endarterectomy (CEA) procedure until the date of hospital discharge, assessed up to 30 days
  Healthcare endpoint : number of days the patient stayed in the hospital stay
Procedure Delay | From the date of patient randomization until the date of carotid artery stenting (CAS) or endarterectomy (CEA) procedure, assessed up to 15 days
  Operational endpoint: number of days between the date at which the patient is randomized and the date at which the carotid artery stenting (CAS) or endarterectomy) is proceeded
Ischemic Events | From 3 days before procedure to 7 days after procedure.
  Clinical endpoint: Incidence of ischemic events among patients with confirmed new lesions on post-procedure DWI MRI (as verified by core lab assessment). The pre-treatment DWI MRI will be performed within 3 days before procedure. The post-treatment DWI MRI will be performed within 7 days after procedure.
Hemorrhage | From 3 days before procedure to 7 days after procedure.
  Imaging endpoint : Hemorrhagic transformation on post-treatment MRI. The pre-treatment DWI MRI will be performed within 3 days before procedure. The post-treatment DWI MRI will be performed within 7 days after procedure.

CONTACTS AND LOCATIONS:
Overall Officials: David Calvet, Professor, Study Director — GHU Sainte-Anne, PARIS; Benjamin GORY, Professor, Study Director — CHU NANCY; Antoine MILLON, Professor, Study Director — Hospices Civils de Lyon
Locations (1):
- Centre hospitalier Sainte-Anne, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with GDPR.